CLINICAL TRIAL: NCT07347535
Title: Non-invasive Assessment of Skeletal Muscle Oxygenation in Athletes and Patients With Peripheral Arterial Disease Using Multispectral Optoacoustic Tomography During Standardized Physical Exercise
Brief Title: Non-invasive MSOT Examination of Muscle Oxygenation in Athletes and PAD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Collaborators: PD Dr. med. Ferdinand Knieling, Department of pediatrics, University of Erlangen-Nürnberg (Unknown)
Responsible Party: Principal Investigator, Ulrich Rother, Senior Consultant, Department of Vascular Surgery, University Hospital Erlangen, University Hospital Erlangen
Other Study IDs: MSOT_SPO2RT
Record Dates: First submitted 2025-12-11; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: PAD - Peripheral Arterial Disease
Keywords: MSOT; PAD; Spiroergometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- PAD - peripheral artery disease: Patients with PAD
  Interventions: Diagnostic Test: MSOT - Multispectral optoacustic tomography; Diagnostic Test: CPET
- Triathletes: very fit subjects, who do triathlon
  Interventions: Diagnostic Test: MSOT - Multispectral optoacustic tomography; Diagnostic Test: CPET
- Strength athletes: Strength athletes and bodybuilders
  Interventions: Diagnostic Test: MSOT - Multispectral optoacustic tomography; Diagnostic Test: CPET
- young, unathletic group: Young, healthy and unathletic subjects between 18 - 40 years
  Interventions: Diagnostic Test: MSOT - Multispectral optoacustic tomography; Diagnostic Test: CPET
- older, unathletic group: older, unathletic and healthy subjects between 55 - 75 years
  Interventions: Diagnostic Test: MSOT - Multispectral optoacustic tomography; Diagnostic Test: CPET
- training PAD Patients
  Interventions: Diagnostic Test: MSOT - Multispectral optoacustic tomography; Diagnostic Test: CPET

INTERVENTIONS:
Diagnostic Test: MSOT - Multispectral optoacustic tomography — MSOT is an advanced imaging technology that combines laser-induced ultrasound and light absorption to visualize biological tissues. By detecting ultrasound waves generated from tissue absorption of multispectral light, MSOT provides high-resolution, real-time images with functional and molecular information. One of its use is in biomedical research and clinical applications to study blood oxygenation and tissue composition, making it valuable for areas such as vascular research. In this study, we aim to utilize MSOT to differentiate between venous, arteriovenous and lymphatic malformations.
Diagnostic Test: CPET — Spiroergometry (also called cardiopulmonary exercise testing, CPET) is a diagnostic test that measures how the heart, lungs, and muscles work together during physical activity. While a person performs exercise treadmill the test records breathing gases (oxygen uptake and carbon dioxide output), ventilation, heart rate, and workload.
  It provides valuable information about aerobic capacity, endurance, and limitations caused by cardiovascular, pulmonary, or metabolic conditions, making it useful in sports medicine, rehabilitation, and clinical diagnostics.

SUMMARY:
The aim of the study is to present the quantitative differences in oxygenated hemoglobin in different cohorts.

This clinical study evaluates whether there is a correlation between measurements using multispectral optoacoustic tomography and the results of spiroergometry in the context of performance diagnostics.

DETAILED DESCRIPTION:
This study aims to investigate the muscle metabolism of athletes (endurance and strength athletes), PAD patients, and healthy control subjects using non-invasive multispectral optoacoustic tomography as part of interval treadmill spiroergometry. The aim is to take a closer look at changes in oxygen supply and muscle metabolism in the various patient groups during the recovery phase. To this end, the individual groups will perform a performance diagnosis on a treadmill spiroergometer, adapted to their respective estimated physical performance (in the case of PAD patients, taking into account the possibilities given by the disease), which will be carried out in the form of a step test. In addition, MSOT measurements will be taken between the individual steps.

The aim of this study is to use MSOT to visualize and compare the muscle perfusion-in particular the proportion of oxygenated and deoxygenated hemoglobin (Hb)-of the various cohorts, as well as to compare it with the diagnostics and methods commonly used to date and identify any advantages. In the future, this could contribute to a better understanding of muscle perfusion, especially in connection with diseases such as PAD or other muscle lesions in sports medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (adults capable of giving consent)
* Capacity to consent. The subjects are able to understand the information provided and give their written consent.
* Belonging to one of the following cohorts:
* Endurance athletes: at least 3× per week ≥ 60 minutes of intensive endurance training (e.g., running, cycling, swimming)
* Strength athletes: at least 3× per week ≥ 60 minutes of intensive strength training without additional endurance training
* Healthy control subjects: less than 2× per week < 30 minutes of physical activity, no known vascular diseases
* PAD patients: diagnosed peripheral arterial occlusive disease in Fontaine stage I or IIa Women of childbearing age with or without contraception may participate, as there are no risks of harm to the fetus.
* Consent to pseudonymized data collection and storage in accordance with the GDPR.

Exclusion Criteria:

* Age over 75 years
* Minors (Age < 18)
* safety concerns on the part of the study physician, e.g., in the case of of: physical, mental or psychiatric illnesses, acute or chronic conditions that could jeopardise safety or data quality
* Taking medications that could affect physical performance or physiological measurements (e.g., heart rate, oxygen uptake).
* Pregnancy with known risks or complications (participation is possible in principle, but subject to individual medical review).
* Refusal to participate or lack of informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include adult participants aged 18 to 75 years, representing different levels of physical activity and vascular health status. A total of approximately 60 participants will be recruited, divided into six cohorts of about ten individuals each.
  Cohort Description:
  * Young endurance athletes (≥ 3 times per week, ≥ 60 minutes per session) Examples: running, cycling, swimming
  * Young strength athletes (≥ 3 times per week, ≥ 60 minutes) No additional endurance training
  * Young healthy controls Less than 2 times per week and < 30 minutes of physical activity No known vascular or muscular diseases
  * Patients with peripheral arterial disease (PAD) Diagnosed with PAD, Fontaine stage I, IIa or IIb
  * Older inactive controls Age above 55 years, no regular physical activity, no pAVK
  * Patients with PAD (Fontaine stage I, IIa or IIb, who participate in structured walking training
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin associated parameters measured via Multispectral optoacoustic Tomography | through study completion, an average of 1 year
  using MSOT
Peak oxygen uptake (VO₂peak): VO₂peak (mL·kg-¹·min-¹) | through study completion, an average of 1 year
  Peak oxygen uptake measured during cardiopulmonary exercise testing (CPET), defined as the highest oxygen uptake achieved during maximal exercise.
Respiratory exchange ratio (RER): RER (VCO₂/VO₂, unitless) | Through study completion, average of 1 year
  Respiratory exchange ratio measured during cardiopulmonary exercise testing (CPET) and calculated as the ratio of carbon dioxide production to oxygen consumption (VCO₂/VO₂).
Minute ventilation: Ventilation (L·min-¹) | Through study completion, average of 1 year
  Minute ventilation measured during cardiopulmonary exercise testing (CPET).
Carbon dioxide production (VCO₂): VCO₂ (mL·min-¹) | Through study completion, average of 1 year
  Carbon dioxide production measured during cardiopulmonary exercise testing (CPET).
Heart rate response to exercise: Heart rate (bpm) | Through study completion, average of 1 year
  Heart rate measured at peak exercise during cardiopulmonary exercise testing (CPET).
Absolute oxygen consumption: VO₂ (mL·min-¹) | Through study completion, average of 1 year
  Oxygen consumption measured during cardiopulmonary exercise testing (CPET).
Anaerobic threshold: HR or workload at AT unit: bpm or km/h | Through study completion, average of 1 year
  Heart rate and workload at anaerobic threshold determined during cardiopulmonary exercise testing (CPET).
Breathing reserve; Percentage (%) | Through study completion (an average of 1 year)
  using CPET Breathing reserve measured during cardiopulmonary exercise testing (CPET) and calculated as the percentage difference between maximal voluntary ventilation and peak exercise ventilation.
Ventilatory equivalent for oxygen (VE/VO₂): Unitless | Through study completion (an average of 1 year)
  Ventilatory equivalent for oxygen measured during cardiopulmonary exercise testing (CPET) and defined as the ratio of minute ventilation to oxygen consumption.
Ventilatory equivalent for carbon dioxide (VE/VCO₂): Unitless | Through study completion (an average of 1 year)
  Ventilatory equivalent for carbon dioxide measured during cardiopulmonary exercise testing (CPET) and defined as the ratio of minute ventilation to carbon dioxide production.